CLINICAL TRIAL: NCT02703636
Title: A 24-week, Open-label, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of Rivastigmine Patch With 1-step Titration in Patients With Mild to Moderate Alzheimer's Disease (MMSE 10 - 23) Switched Directly From Holinesterase Inhibitors (Donepezil, Galantamine)
Brief Title: NextStep:Study to Evaluate Safety,Efficacy & Tolerability of Rivastigmine Patch in Mild to Moderate Alzheimer's Patients.
Acronym: ENA1stepswitch
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENA713DJP02
Record Dates: First submitted 2016-02-26; First posted 2016-03-09 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Mild to Moderate Alzheimer's Disease
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Rivastigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rivastigmine Patch (Other): Alzheimer's disease patient who is applicable to 1 step titration method (initial loading dose is a rivastigmine patch 9.0 mg/day and will be up-titrated after 4 weeks to reach the maintenance dose of 18 mg/day). Rivastigmine patch is a marketed drug, therefore the dose, dose regimen and titration scheme are in accordance with product label.
  Interventions: Drug: Rivastigmine Patch

INTERVENTIONS:
Drug: Rivastigmine Patch — Alzheimer's disease patient who is applicable to 1 step titration method (initial loading dose is a rivastigmine patch 9.0 mg/day and will be up-titrated after 4 weeks to reach the maintenance dose of 18 mg/day). Rivastigmine patch is a marketed drug, therefore the dose, dose regimen and titration scheme are in accordance with product label.
  Other Names: rivastigmine

SUMMARY:
To evaluate the efficacy of rivastigmine patch with 1-step titration on cognitive function measured as change from baseline to week 24 in the total score of Mini-Mental State Examination (MMSE) in mild to moderate Alzheimer's disease (AD) patients who failed to benefit from other cholinesterase inhibitors (ChEIs).

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient status at baseline.
2. Males, and females not of child-bearing potential (surgically sterile, or one year or more from last menses).
3. A diagnosis of dementia of the Alzheimer's type according to the DSM-IV criteria.
4. A clinical diagnosis of probable AD according to National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
5. Brain scan (magnetic resonance imaging [MRI], or computed tomography [CT]) were met diagnosis criteria conducted within 3 years prior to baseline.
6. Positron emission tomography (PET) or single photon emission computed tomography (SPECT) was met diagnosis criteria conducted within 3 years prior to baseline visit, as long as in the past a brain scan (MRI or CT) also was met.
7. MMSE score of ≥ 10 and ≤ 23 at screening and baseline.
8. Patients are currently on the oral monotherapy (donepezil, 5 mg), or galantamine (16-24 mg) for 4 weeks prior to baseline visit.
9. Patients who failed to receive enough treatment benefit from the previous treatment can be defined if the patients meet at least one of following conditions at screening and baseline (multiple choices allowed)
10. Patients who declined ≥ 2 points of MMSE despite of treatment of other oral Cholinesterase (ChE) inhibitors within initial 3-month and continued to show insufficient treatment effect until at baseline.
11. During 6 months prior to screening visit, patients who declined ≥2 points of MMSE with other oral ChE inhibitors and continued to show insufficient treatment effect until at baseline.
12. Patients who show marked worsening of BPSD, or ADL (can be defined by 1 state progression of FAST) judged by a physician despite of treatment of other oral ChE inhibitors in initial 3-month or last 6-month with other oral ChE inhibitors
13. Patients having difficulties being treated orally with ChEIs (donepezil or galantamine) by physician's judgement.
14. Poor compliance or adverse event except GI symptoms
15. Patients with swallowing difficulties.

Exclusion Criteria:

1. Any medical or neurological condition other than AD that could explain the patient's dementia (e.g., abnormal thyroid function tests, vitamin B12 or folate deficiency, posttraumatic conditions, syphilis, head injury, Huntington's disease, Parkinson's disease, subdural hematoma, normal pressure hydrocephalus, brain tumor) at baseline
2. Any other DSM-IV Axis 1 diagnosis that may interfere with the evaluation of the patient's response to study medication, including other primary neurodegenerative dementia, schizophrenia, or bipolar disorder
3. An advanced, severe, progressive, or unstable disease of any type that may interfere with efficacy and safety assessments or put the patient at special risk
4. Current diagnosis of an active skin lesion/disorder
5. Patients with a history of hypersensitivity to any ingredients of rivastigmine or carbamate derivatives
6. Each patient will be required to have a primary caregiver willing to accept responsibility for supervising treatment, assessing the patient's condition throughout the study, and for providing input into efficacy assessments.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- Japan (18):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Aizu-Wakamatsu, Fukushima
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Kochi, Kochi
  - Novartis Investigative Site, Sanjō, Niigata
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Kasukabe, Saitama
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Fuji, Shizuoka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Suginami Ku, Tokyo
  - Novartis Investigative Site, Okayama

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The full analysis set (FAS) included all patients who received at least one dose of study treatment and had at least a baseline and any post-baseline assessment on treatment.
Pre-assignment Details: In total, 147 patients were screened for the study. 129 completed screening and 18 discontinued from screening. 118 patients were enrolled and the remaining 11 patients discontinued at baseline.
  All 118 enrolled patients received study treatment. 102 completed the study and 16 discontinued
Groups:
- Rivastigmine Patch: Alzheimer's disease patient who is applicable to 1 step titration method (initial loading dose is a rivastigmine patch 9.0 mg/day and was up-titrated after 4 weeks to reach the maintenance dose of 18 mg/day). Rivastigmine patch is a marketed drug, therefore the dose, dose regimen and titration scheme are in accordance with product label.
Period: Overall Study
Arm/Group | Rivastigmine Patch
Started | 118
Completed | 102
Not Completed | 16
Not completed — Adverse Event | 14
Not completed — Study stopped by sponsor | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: FAS
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.4 (6.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 117
  Caucasian | 1

OUTCOME MEASURES:

1. Primary Outcome: MMSE Total Score: Change From Baseline to Week 8 and Week 24 (Full Analysis Set)
Description: Evaluation of the efficacy of rivastigmine patch with 1-step titration on cognitive function measured as change from baseline to week 24 in the total score of MMSE in mild to moderate Alzheimer's disease (AD) patients who failed to benefit from other cholinesterase inhibitors (ChEIs)
  The MMSE is a screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); the total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement from baseline.
  Abbreviated Scale title: Mini Mental State Evaluation Minimum Score: 0 Maximum score: 30 Higher score indicated better cognitive function
Time Frame: baseline, weeks 8 and 24
Population: The full analysis set (FAS) included all patients who received at least one dose of study treatment and had at least a baseline and any post-baseline assessment on treatment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 118
scores on a scale
  baseline | 17.33 (3.80)
  change at week 8: number analyzed (Participants) | 117
  change at week 8 | 0.29 (2.17)
  change at week 24: number analyzed (Participants) | 102
  change at week 24 | -0.36 (2.64)
Statistical Analysis 1: Comparison: Rivastigmine Patch; Test type: Other — The MMRM model contained visit as a fixed effect, baseline MMSE score as a covariate and patient as a random effect; p = 0.1750, t-test, 2 sided; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.87 to 0.16], Standard Error of Mean 0.259 — change at week 24

2. Secondary Outcome: MMSE Total Score: Change From Baseline to Week 8 and Week 24
Description: Evaluation of the safety, tolerability of rivastigmine patch with 1-step titration for up to 24 weeks.
  Per Protocol, The MMSE is a brief, practical screening test for cognitive dysfunction. The MMSE consists of 2 parts: language (time orientation, registration and attention) and performance (recall, response to written/verbal commands, writing ability and reproduction of complex polygons), and the total possible score is 30. Lower score indicates more severe impairment. It is the most common and simple cognitive scale for Alzheimer's disease.
  Unabbreviated Scale : MMSE - Mini Mental State Evaluation:
  Minimum values - 0 Maximum value - 30 Higher Value means a better outcome
  Positive change score from baseline indicates improvement in cognitive function
Time Frame: baseline, weeks 8 and 24
Population: Per Protocol Set (PPS): The per protocol set includes all patients in the FAS who had only 1 step titration without any major deviations from the protocol procedures
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 118
scores on a scale
  baseline: number analyzed (Participants) | 112
  baseline | 17.24 (3.84)
  week 8: number analyzed (Participants) | 112
  week 8 | 0.33 (2.19)
  week 24: number analyzed (Participants) | 98
  week 24 | -0.32 (2.63)

3. Secondary Outcome: Change From Baseline to Week 8 in Mini-Mental State Examination (MMSE) Total Score
Description: Evaluation of the efficacy of rivastigmine patch with 1-step titration measured as the MMSE score at week 8 for patients who had 1-step titration
  MMSE total score: change from baseline to Week 8 and Week 24 for patients who had 1-step titration
  Unabbreviated Scale : MMSE - Mini Mental State Evaluation:
  Minimum values - 0 Maximum value - 30 Higher Value means a better outcome
  Positive change score from baseline indicates better outcome
Time Frame: baseline and week 8
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 114
scores on a scale
  baseline | 17.25 (3.82)
  week 8 | 0.31 (2.18)

4. Secondary Outcome: Change in Neuropsychiatric Inventory - 10 Item (NPI-10) Score From Baseline to Week 8 and Week 24
Description: Evaluation of the efficacy of rivastigmine patch with 1-step titration measured as the Neuropsychiatric Inventory - 10 Item (NPI-10) score at week 8 and week 24.
  Per protocol, Neuropsychiatric The NPI-10 total score is a sum of the 10 items, where the score for a domain is defined as the product of frequency (range: 1-4) and severity (range: 1-3). Each domain has a maximum score of 12 and all domains are equally weighted for the total score (thus the range for the total score is 0 to 120).
  A higher score indicates more severe impairment.
  Neuropsychiatry Inventory - 10 Minimum Score = 0 Maximum Score = 120
  Higher Score indicates worse outcome
Time Frame: baseline, week 8, week 24
Population: FAS The number of participants analysed per row differs from overall number of participants because this is based on available data and patient continuation/discontinuation during that respective study period.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 118
scores on a scale
  baseline | 11.43 (11.15)
  week 8: number analyzed (Participants) | 116
  week 8 | -1.81 (8.81)
  week 24: number analyzed (Participants) | 102
  week 24 | -0.89 (11.10)

5. Secondary Outcome: Change in QOL-AD Score From Baseline to Week 24
Description: Evaluation of the efficacy of rivastigmine patch with 1-step titration measured as QOL-AD score at week 24.
  Unabbreviated Scale Name: Quality of Life - Alzheimer's Disease Minimum Score = 13 Maximum Score = 52
  Higher value indicates a better outcome
  QOL-AD is a 13-item questionnaire to assess the quality of life of Alzheimer's patients from the perspectives of patients and their caregivers. It covers several aspects, for example, the perception of health status, mood, functional capacity, personal relationships and leisure, financial situation, and life as a whole. Each item is quantified using a Likert scale with score one classified as poor, and score four as excellent where total scores range from 13 to 52. A lower score indicates more severe impairment.
Time Frame: baseline and week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 118
scores on a scale
  baseline - Patient's assessment | 34.37 (5.78)
  week 24 - Patient's assessment: number analyzed (Participants) | 102
  week 24 - Patient's assessment | -0.34 (5.32)
  baseline - Caregiver's assessment | 28.75 (5.74)
  week 24 - Caregiver's assessment: number analyzed (Participants) | 103
  week 24 - Caregiver's assessment | -0.16 (5.42)

6. Secondary Outcome: Change in J-CGIC Score From Baseline and at Week 24
Description: Evaluation of the efficacy of rivastigmine patch with 1-step titration measured as the The Japanese-Clinical Global Impression of Change (J-CGIC) score at baseline and week 24
  J-CGIC is a 7-grade investigator's impression scale: 1. Markedly improved, 2. Improved, 3. Slightly improved, 4. No change, 5. Slightly aggravated, 6. Aggravated, 7. Markedly aggravated
  At week 24, 103 patients had available data
  Total score is in the 0 to 56 range. Higher score means more severe impairment.
  Unabbreviated scale title: Japanese -Cinical Global Impression of Change Minimum Score - 1 Maximum Score - 7
Time Frame: baseline and week 24
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 103
Participants
  Patients without worsening, total | 91
  Patients with improvement | 48
  Patients with worsening, total | 12
  Markedly improved | 3
  Improved | 6
  Slightly improved | 39
  No change | 43
  Slightly aggravated | 11
  Aggravated | 1
  Markedly aggravated | 0
  Unassessable | 0

7. Secondary Outcome: Change in as Modified Crichton Scale Score From Baseline to Week 4, 8, 16 and 24
Description: Evaluation of the efficacy of rivastigmine patch with 1-step titration measured as Modified Crichton Scale score week 4, week 8, week 16, and week 24.
  Modified Crichton Scale that assess basic activation of daily living, communication functions, and quality of life The following 7 items will be evaluated by caregiver. Total score is in the 0 to 56 range. Higher score means more severe impairment.
  Unabbreviated Scale Title: Modified Crichton scale Minimum score = 0 Maximum Score = 56 Higher score indicates worse outcome
Time Frame: baseline, weeks 4, 8, 16, 24
Population: FAS
  The number of participants analysed per row (modified crichton scale) differs from overall number of participants because this is based on available data and patient continuation/discontinuation during that respective study period.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 118
scores on a scale
  baseline | 18.38 (9.41)
  week 4: number analyzed (Participants) | 117
  week 4 | -0.41 (5.44)
  week 8: number analyzed (Participants) | 116
  week 8 | -0.55 (6.58)
  week 16: number analyzed (Participants) | 108
  week 16 | 1.04 (6.94)
  week 24: number analyzed (Participants) | 103
  week 24 | 2.23 (6.69)

8. Secondary Outcome: Formulation Usability Questionnaire Form Score up to Week 24
Description: Evaluation of the formulation usability of rivastigmine patch for up to 24 weeks as measured by the formulation usability questionnaire answered by caregiver.
  The Formulation usability preference questionnaire had been used to compare the previous oral AD drugs versus the patch The caregiver selects one of the following answers (1. Very easy to use, 2. Easy to use, 3. No change, 4. Not easy to use, 5. Not easy to use at all, 6. Unknown).
  This questionnaire data is used to assess if the usability of rivastigmine patch was preferred by the majority (> 50%) of AD patient caregivers or not.
  Unabbreviated Questionnaire title:
  Formulation Usability questionnaire Minimum Score = 1 Maximum Score = 6
  A higher score indicates its not easy to use and worse outcome.
Time Frame: Up to week 24
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Rivastigmine Patch
Number analyzed (Participants) | 117
Participants
  Very easy to use | 38
  Easy to use | 26
  No change | 12
  Not easy to use | 36
  Not easy to use at all | 5

ADVERSE EVENTS:
Time Frame: up to week 24
Groups:
- Exelon/Rivastigmine Patch: Alzheimer's disease patient who is applicable to 1 step titration method (initial loading dose is a rivastigmine patch 9.0 mg/day and was up-titrated after 4 weeks to reach the maintenance dose of 18 mg/day). Rivastigmine patch is a marketed drug, therefore the dose, dose regimen and titration scheme are in accordance with product label.
Arm/Group | Exelon/Rivastigmine Patch
All-Cause Mortality (participants affected / at risk) | 0/118
Serious Adverse Events (participants affected / at risk) | 5/118
Other Adverse Events (participants affected / at risk) | 57/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exelon/Rivastigmine Patch (N=118)
Ileus (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exelon/Rivastigmine Patch (N=118)
Application site erythema (General disorders) | 9
Application site pruritus (General disorders) | 10
Nasopharyngitis (Infections and infestations) | 12
Dermatitis contact (Skin and subcutaneous tissue disorders) | 18
Erythema (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-08-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT02703636/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT02703636/SAP_001.pdf